CLINICAL TRIAL: NCT00384163
Title: Adult Pulmonary Valve Replacement: A Simple and Reproducible Technique
Status: Terminated | Type: Observational
Why Stopped: sufficient data collected
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Brian Kogon, Associate Professor of Surgery, Emory University
Other Study IDs: 0453-2006
Record Dates: First submitted 2006-10-03; First posted 2006-10-05 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Disorders
Keywords: cardiac; adult; PVR
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Pulmonary valve replacement in the adult population is an uncommon operation. The majority of native valve pathology in adults involves the mitral, aortic, and occasionally tricuspid valves. On the other hand, right ventricular outflow tract and pulmonary valve disease is quite common in children, especially with tetralogy of fallot, truncus arteriosus, pulmonary atresia/ventricular septal defect, and double outlet right ventricle. Unfortunately, right ventricular pathology often develops in adulthood as a result of pulmonary insufficiency or pulmonary stenosis created by previous childhood operations. Without the valve size constraints present at prior operations, these patients can be well-served by the placement of adult-sized bioprosthetic valves. There are limited descriptions in the adult cardiac literature of the actual technique of pulmonary valve replacement. We present our current technique and the pitfalls encountered when performing pulmonary valve replacement in adults.

DETAILED DESCRIPTION:
This will be primarily a technique paper. The only clinical data points I am interested in are the presence of pulmonary stenosis, pulmonary insufficiency or perivalvular leak on the initial post-operative echocardiogram. I estimate reviewing 50 patients' charts dated March 22.2003 through and including March 22.2006 at Emory Hospital .

Primary Aim: Present an effective technique for pulmonary valve replacement

Secondary Aim: Present our excellent technical results of PVR in our adult congenital patients

ELIGIBILITY:
Inclusion Criteria:

* Adults undergoing pulmonary valve replacement
* at Emory Hospital
* between 3.22.03 amd 3.22.06

Exclusion Criteria:

* those charts that do not fall under inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2007-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Kogon, MD, Principal Investigator — Emory University SOM
Locations (1):
- Emory University, Atlanta, Georgia, United States